CLINICAL TRIAL: NCT01482936
Title: A Single Dose PK Study of Oxycodone Hydrochloride Injection 2.5, 5, and 10mg in Chinese Patients With Cancer Pain or Post-operation Patients
Brief Title: Pharmacokinetic (PK) Study of OxyNorm Injections in Chinese Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXYI09-CN-101
Record Dates: First submitted 2011-11-17; First posted 2011-12-01 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone (OxyNorm®) Injection (Experimental): The subjects will be randomized to receive a single dose of OxyNorm® 2.5, 5, and 10mg
  Interventions: Drug: Oxycodone (OxyNorm®) Injection

INTERVENTIONS:
Drug: Oxycodone (OxyNorm®) Injection — The subjects will be randomized to receive a single dose of OxyNorm® 2.5, 5, and 10mg.The plasma concentration will be analyzed to determine the following pharmacokinetic parameters:AUC0-t:ug•hr/L-Area under the plasma concentration-time curve frame: predose,0,2min,5min,10min,15min,30min,45min,1hr,1.5hr,2hr,3hr,4hr,6hr,8hr,12hr, 24hr post-dose.AUC0-inf:ug•hr/L-Area under the plasma concentration-time curve extrapolated to infinity. Cmax: ug/L-Maximum observed plasma concentration of oxycodone and noroxycodone.Tmax: hrs-time at which Cmax is first observed. t½: Apparent half life of oxycodone elimination.
  Other Names: OxyNorm®

SUMMARY:
This is a single center, open label, randomized, parallel group single dose intravenous (i.v.) administration study. The subjects will be randomized to receive a single dose of OxyNorm® 2.5, 5, and 10mg.

DETAILED DESCRIPTION:
After up to 7 days screening period, Eligible Patients will be randomized to 1 of 3 groups, and begin treatment with single dose of OxyNorm® 2.5,5, and 10mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumor pain / postoperative pain, or subjects with pain caused by other diseases;
* Patients aged >30 to ≤ 60 years;
* Body weight ≥ 45kg, and BMI range ≥19, <24;
* Karnofsky score ≥ 70;
* Expected survival is above 3 months;
* The results of liver function and kidney tests must meet the following criteria:ALT、AST is within the upper limit of normal value ranges by a factor 2, and TB、BUN、Cr is within the upper limit of normal value ranges by a factor 1.25;
* The electrocardiogram examination results are normal;
* Patients must have given a written informed consent prior to this trial, and have the capability to complete every required test.

Exclusion Criteria:

* Have hypersensitivity history to any opioids;
* Have known hypersensitivity to any of compositions of the study drugs;
* Patients who are likely to have paralytic ileus or acute abdomen or to perform an operation on abdominal region；
* Patients with respiratory depression, cor pulmonary, or chronic bronchial asthma;
* Patient unable to stop taking monoamine oxidase inhibitor during this trial period or time lapses less than 2 weeks since drug withdrawal;
* Patients with hypercarbia;
* Patients with biliary tract diseases, pancreatitis, prostatic hypertrophy, or corticoadrenal insufficiency;
* Patients with alcoholism or drug abuse history;
* Positive ant-HIV or syphilis antibody test result;
* Urine screening before study is positive for the opioids, barbiturates, amphetamines, cocaine metabolites, methadone, diazepam and cannabinoids;
* Donated 400 mL or more of blood or blood products within 3 months prior to the start of the study, or donated 200 mL or more of blood or blood products within one month prior to the start of the study.
* Subjects who participated in a clinical research study within two months of study entry.
* Patients who are currently taking opioids.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) concentrations of oxycodone hydrochloride injection at various time points: predose, 0min, 2min, 5min, 10min, 15min, 30min, 45min, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24hr post dose. | 2 days
  Plasma concentrations of oxycodone and Noroxycodone and Oxymorphone will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mundipharma China Ltd., Study Chair — Mundipharma China Ltd.
Locations (1):
- Investigational Site: Affiliated Hospital to Academy of Military Medical Science of China People's Liberation Army, Beijing, China